CLINICAL TRIAL: NCT05444985
Title: Post-operative Analgesic Effects of Bilateral External Oblique Intercostal Block in Laparoscopic Cholecystectomy Surgeries.
Brief Title: Postoperative Analgesic Effects of Bilateral External Oblique Intercostal Block in Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HATICE55
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Analgesia; Pain, Postoperative
Keywords: External oblique intercostal block; Pain management
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Pain Management

STUDY DESIGN:
Intervention Model Description: One interventional group and one control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The anesthetist who will perform the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another anesthetist blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Oblique Intercostal Block Group (Experimental): While patients are still under general anesthesia, external oblique intercostal block (EOIB) will be performed bilaterally according to appropriate asepsis/antisepsis rules before awakening.
  Interventions: Other: Pain Management
- Control (Active Comparator): Patients in the control group will not have any intervention concerning regional anesthesia.
  Interventions: Other: Pain Management

INTERVENTIONS:
Other: Pain Management — Regional anesthetic techniques for peri-operative pain management after surgery.

SUMMARY:
The aim of our study is to reduce postoperative pain by performing external oblique intercostal block in L/S cholecystectomy surgeries. Our main goal is to provide well managed post-operative analgesia.

DETAILED DESCRIPTION:
The patients will be divided into two groups and general anesthesia will be applied to all of them. There will be no regional anesthetic technique to be performed, on the other hand, external oblique intercostal nerve block will be applied to patients in the other group before the patients are extubated. Study randomization is done with computer-generated randomization codes (computer-generated) by a physician who will not participate in patient follow-up. Interfascial plane block (external oblique intercostal block) will be given to the anesthesiologist in a sealed envelope by an independent assistant staff outside the study, the patient will not know which block is applied. The anesthetist who made the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another anesthetist blinded to the study.

For the standardization, the block procedure will be performed by an experienced anesthesiologist who has performed at least 20 previous successful and uncomplicated procedures.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m²
* Patients with ASA scores I and II

Exclusion Criteria:

* Patients who do not want to be included in the study
* Psychiatric and neurological disease with blurred consciousness
* Patients with ASA > 3
* BMI > 35 kg/m²
* Abnormality in coagulation parameters
* History of allergy to local anesthetic drugs
* Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Contramal consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
NRS scores | At 1,3, 6, 12, 18, 24 hours
  NRS scores in the first 24 hours after surgery
Quality of recovery | 24 hours
  QR15 scores
Nausea and vomiting | At 1,3, 6, 12, 18, 24 hours
  Nausea and vomiting scores in the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Kusderci, M.D., Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No